CLINICAL TRIAL: NCT06542172
Title: Impact of Low-fat and Full-fat Milk on Lipids and Cardiac Function in Patients With Coronary Artery Disease: A Randomized Controlled Trial
Brief Title: Impact of Low-fat and Full-fat Milk on Lipids and Cardiac Function in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Rong Wang, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: low-fat and full-fat milk
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — CD36 Antigens; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 500 mL/day of low-fat milk (fat <1.5%) (Experimental): All milk is provided by the Inner Mongolia Yili Industrial Group Limited by Share Ltd (Inner Mongolia, China).
  Interventions: Dietary Supplement: 500 mL/day of low-fat milk (fat <1.5%) for 12 weeks
- 500 mL/day of full-fat milk from corn-fed cows (fat >3.8%) (Experimental): All milk is provided by the Inner Mongolia Yili Industrial Group Limited by Share Ltd (Inner Mongolia, China).
  Interventions: Dietary Supplement: 500 mL/day of full-fat milk from corn-fed cows (fat >3.8%) for 12 weeks
- 500 mL/day of full-fat milk from grass-fed cows (fat >3.8%) (Experimental): All milk is provided by the Inner Mongolia Yili Industrial Group Limited by Share Ltd (Inner Mongolia, China).
  Interventions: Dietary Supplement: 500 mL/day of full-fat milk from grass-fed cows (fat >3.8%) for 12 weeks

INTERVENTIONS:
Dietary Supplement: 500 mL/day of full-fat milk from corn-fed cows (fat >3.8%) for 12 weeks — All milk is provided by the Inner Mongolia Yili Industrial Group Limited by Share Ltd (Inner Mongolia, China).
  Arms: 500 mL/day of full-fat milk from corn-fed cows (fat >3.8%)
Dietary Supplement: 500 mL/day of full-fat milk from grass-fed cows (fat >3.8%) for 12 weeks — All milk is provided by the Inner Mongolia Yili Industrial Group Limited by Share Ltd (Inner Mongolia, China).
  Arms: 500 mL/day of full-fat milk from grass-fed cows (fat >3.8%)
Dietary Supplement: 500 mL/day of low-fat milk (fat <1.5%) for 12 weeks — All milk is provided by the Inner Mongolia Yili Industrial Group Limited by Share Ltd (Inner Mongolia, China).
  Arms: 500 mL/day of low-fat milk (fat <1.5%)

SUMMARY:
This trial aimed to investigate the effects of low-fat and full-fat milk on patients with coronary artery disease (CAD).

DETAILED DESCRIPTION:
The effects of low-fat and full-fat milk on lipid profiles and sphingolipid profiles in CAD patients are not well understood. In addition, milk intake is at a low level in the Chinese population compared with developed countries. Therefore, we aimed to conduct a randomized controlled trial to investigate the effects of low-fat and full-fat milk on lipid profiles, sphingolipid profiles, and cardiac performance in Chinese CAD patients.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients with CAD

Exclusion Criteria:

(1) patients <18 years of age; (2) patients with systemic active infection; (3) patients with severe hepatic and renal dysfunction [alanine aminotransferase (ALT) > 135mmol/L, creatinine > 200umol/L), or chronic lung disease; (4) patients with a life expectancy ≤ 6 months due to bleeding tendency and hematological diseases, malignant tumors, and end-stage diseases; (5) patients with valvular heart disease or left ventricular aneurysm who needed simultaneous surgeries; (6) patients with cerebrovascular disease (cerebral infarction or cerebral hemorrhage within 6 months before enrollment); (7) patients who enrolled in other drug intervention trials; (8) patients who received emergency percutaneous coronary intervention (PCI); and (9) patients who reported intolerance to lactose.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
differences in lipids, sphingolipids, and cardiac function between the three groups after 12 weeks of intervention | after 12 weeks of intervention
  The lipids contain total cholesterol, triglycerides, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), small dense LDL (sd LDL), large buoyant LDL (lb LDL), phospholipids, apolipoprotein A Ⅰ (apoA Ⅰ), apolipoprotein B (apoB), and lipoprotein (a). Sphingomyelins (C16:0, C20:0, C20.1:0, C22:0, C24.1:0) as well as their metabolites such as ceramides (C16:0, C18:0, C18.1:0, C20:0, C20.1:0, C22:0, C24:0, C24.1:0), sphingosine, and sphingosine 1-phosphate, were also measured.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Wang, MD, Principal Investigator — Chinese PLA General Hospital
Locations (7):
- China (7):
  - Beijing Chaoyang Hospital Affiliated to Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - Dongzhimen Hospital, Beijing
  - The Third Military Medical University of the Chinese people's Liberation Army, Chongqing
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - Nanjing First Hospital, Nanjing
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No